CLINICAL TRIAL: NCT07350577
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety Tolerability, Pharmacokinetics, and Pharmacosymics of Single Ascending Doses of Intravenously Administerted ALTB-268 in Healthy Participants
Brief Title: Evaluate the Safety, Tolerability, PK and PD of SAD of Intravenously Adminsterted ALTB-268 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AltruBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ALTB-268-102
Record Dates: First submitted 2025-12-01; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Biological: ALTB-268 (Experimental): Intravenously administered
  Interventions: Biological: ALTB-268
- Placebo (Saline solution) (Placebo Comparator): Intravenously Administered
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ALTB-268 — monoclonal antibody
  Arms: Biological: ALTB-268
Other: Placebo — Saline solution
  Arms: Placebo (Saline solution)

SUMMARY:
This study with ALTB-268 will determine the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending doses of intravenously administrated ALTB-268 in healthy participants.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, single ascending dose (SAD) study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of intravenously administered ALTB-268 in healthy participants. Approximately 24 healthy participants will be recruited.

The primary objective is to evalute the safety and tolerability of intravenous infusion of SAD in healthy participants. The secondary objectives are (1) to characterize the PK profile of ALTB-268 in plasma following single IV doses in healthy participants, and (2) to assess the PD of ALTB-268 following single IV doses in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥18 and ≤55 years of age, with body mass index (BMI) >18.5 and <32.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic diseases.
3. Female participants of non-childbearing potential must be:

   1. post-menopausal (spontaneous amenorrhea for at least 12 consecutive months prior to dosing) with confirmation by documented follicle- stimulating hormone (FSH) levels ≥40 mIU/mL; or
   2. surgically sterile (bilateral oophorectomy, bilateral salpingectomy, hysterectomy, or bilateral tubal ligation) at least 3 months prior to dosing.
4. Able to understand the study procedures, agree to comply with all study visits, procedures, and restrictions, agree to comply with the prescribed dosage regimens and communicate to study personnel about AEs and concomitant medication use, and provide signed informed consent to participate in the study.

Exclusion Criteria:

1. Any clinically significant abnormal finding at physical examination at screening and/or Day -1.
2. Clinically significant abnormal laboratory test results at screening and/or Day -1; or positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody, or QuantiFERON®-TB test at screening.
3. Any history of suicidal ideation as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the C-SSRS completed at screening, or any history of suicide attempts.
4. Any history of clinical depression.
5. C-SSRS score at Day -1 (baseline) above Type 1 ideation.
6. PHQ-8 total score ≥5 at screening and/or Day -1 (baseline).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ALTB-268 following intravenous (IV) infusion in healthy participants - Adverse Events | Through study completion, up to day 71 of the study
  - Numbers of participants with adverse events (AEs): seriousness, severity, relationship to the investigational products, outcome, duration, and management
To evaluate the safety and tolerability of ALTB-268 following intravenous (IV) infusion in healthy participants - Infusion Site Assessments | Through study completion, up to day 71 of the study
  - Infusion site assessments, the extent of local reaction at the infusion site will be graded using the scores described below; a global severity rating for infusion site reactions will be included in the assessment of AEs.
  Infusion Site Reaction Score:
  None: No reaction; Mild: Tenderness with or without associated symptoms; Moderate: Pain; lipodystrophy; edema; phlebitis; Severe: Ulceration or necrosis; severe tissue damage; operative intervention indicated.
To evaluate the safety and tolerability of ALTB-268 following intravenous (IV) infusion in healthy participants - C-SSRS | Through study completion, up to day 71 of the study
  - Columbia suicidality severity rating scale (C-SSRS) is a suicidal ideation and behavior rating scale to evaluate suicide risk.
To evaluate the safety and tolerability of ALTB-268 following intravenous (IV) infusion in healthy participants - PHQ-8 | Through study completion, up to day 71 of the study
  - Patient Health Questionnaire-8 (PHQ-8) depression scale is used for depression screening and severity.
To evaluate the safety and tolerability of ALTB-268 following intravenous (IV) infusion in healthy participants - Clinical Laboratory Test | Through study completion, up to day 71 of the study
  - Clinical laboratory test results, including white blood cell, lymphocyte and neutrophail (cell counts/ul).

SECONDARY OUTCOMES:
Pharmacokinetic (PK) of ALTB-268 AUC | Through study completion, up to day 71 of the study
  * AUC0-t, area under the concentration-time curve from time 0 to t hours
  * AUC0-inf, area under the concentration-time curve from time 0 to infinity
Pharmacokinetic (PK) of ALTB-268 Cmax | Through study completion, up to day 71 of the study
  Mmaximum concentration (Cmax)
Pharmacokinetic (PK) of ALTB-268 Tmax | Through study completion, up to day 71 of the study
  Time to reach Cmax (Tmax)
Pharmacokinetic (PK) of ALTB-268 T½ | Through study completion, up to day 71 of the study
  Terminal half-life (T½)
Pharmacokinetic (PK) of ALTB-268 CL | Through study completion, up to day 71 of the study
  Total body clearance (CL)
Pharmacokinetic (PK) of ALTB-268 Vz | Through study completion, up to day 71 of the study
  Volume of distribution (Vz)
Pharmacokinetic (PK) of ALTB-268 Vss | Through study completion, up to day 71 of the study
  Steady-state volume of distribution (Vss)
Pharmacodynamics (PD) of ALTB-268 following single IV doses in healthy participants. | Through study completion, up to day 71 of the study
  Levels of free soluble P-selectin glycoprotein ligand-1 (sPSGL-1) in plasma.
Immunogenicity of ALTB-268 in plasma following single IV doses in healthy participants | Through study completion, up to day 71 of the study
  Incidence and level of anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health Clinical Research Services, LLC, Miami, Florida, United States